CLINICAL TRIAL: NCT07116551
Title: Abbott BE TAVI Early Feasibility Study: Early Feasibility Study (EFS) of Abbott's Balloon-expandable (BE) TAVI System for the Treatment of Severe, Symptomatic Aortic Stenosis
Brief Title: Early Feasibility Study (EFS) of Abbott's Balloon-expandable (BE) TAVI System for the Treatment of Severe, Symptomatic Aortic Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ABT-CIP-10541
Record Dates: First submitted 2025-07-22; First posted 2025-08-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Symptomatic Severe Aortic Stenosis
Keywords: Balloon Expandable TAVI; TAVI; Treatment of patient with symptomatic severe aortic valve stenosis; aortic stenosis; cardiovascular disease
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BE TAVI System (Experimental): BE TAVI System
  Interventions: Device: Abbott BE TAVI System

INTERVENTIONS:
Device: Abbott BE TAVI System — Abbott BE TAVI System

SUMMARY:
The purpose of this study is to evaluate the safety and functionality of Abbott's BE TAVI system for the treatment of patients with symptomatic severe aortic valve stenosis.

DETAILED DESCRIPTION:
The EFS will evaluate the safety and functionality of Abbott's BE TAVI system for the treatment of patients with symptomatic severe aortic valve stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject is able and willing to return for required follow-up visits and assessments
* Degenerative severe aortic valve stenosis of the native aortic valve with echo-derived criteria

Exclusion Criteria:

* Pregnant or nursing subjects
* Life expectancy for a condition other than aortic stenosis is less than 2 years
* Presence of other anatomic or comorbid conditions
* Incapacitated individuals
* Evidence of an acute myocardial infarction
* Untreated clinically significant coronary artery disease requiring revascularization
* Liver failure
* Severe mitral regurgitation or severe mitral stenosis
* etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-10-30 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Technical success | From start of procedure up to end of procedure
  Successful access, delivery of the Abbott BE TAVI valve, and retrieval of the delivery system.
Device success | 30 days
  Intended performance of the valve

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Oza, Study Director — Abbott Structural Heart
Locations (5):
- United States (4):
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Columbia University Medical Center/New York-Presbyterian, New York, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
- Clinique Pasteur Toulouse, Toulouse, Midpyre, France